CLINICAL TRIAL: NCT06493461
Title: Phase 1b, Multicenter, Open-Label, Multiple Ascending Dose Study Assessing the Pharmacokinetics, Safety, Pharmacodynamics, and Efficacy of HS135 Added to Background Pulmonary Arterial Hypertension (PAH) Therapy
Brief Title: A Study of HS135 for the Treatment of Pulmonary Arterial Hypertension in Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: 35Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS135-002
Record Dates: First submitted 2024-06-28; First posted 2024-07-10 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HS135 (Experimental): Subcutaneous Injection
  Interventions: Biological: HS135

INTERVENTIONS:
Biological: HS135 — HS135 is dosed subcutaneously

SUMMARY:
A Study of HS135 for the Treatment of Pulmonary Arterial Hypertension in Adults

DETAILED DESCRIPTION:
Phase 1b, Multicenter, Open-Label, Multiple Ascending Dose Study Assessing the Pharmacokinetics, Safety, Pharmacodynamics, and Efficacy of HS135 Added to Background Pulmonary Arterial Hypertension (PAH) Therapy

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, 18 years of age and older.
2. Body Mass Index (BMI) 18.5 and 40 kg/m2 and body weight at or below 120 kg
3. Documented diagnostic RHC at any time prior to screening.
4. Diagnosis of WHO PAH Group 1.
5. Symptomatic PAH classified as WHO FC II to IV.
6. Baseline RHC performed during the Screening Period documenting a minimum PVR of ≥ 5 Wood units (WU) or ≥ 400 dyn・sec・cm-5 and a pulmonary artery wedge pressure (PAWP) of ≤ 15 mmHg.
7. On stable doses of at least 2 background PAH therapies.

Exclusion Criteria:

1. Left ventricular ejection fraction < 50% at screening.
2. Any symptomatic coronary disease events within 6 months of the screening visit.
3. Uncontrolled systemic hypertension.
4. History of restrictive, constrictive or congestive cardiomyopathy.
5. History of atrial septostomy.
6. Patients who have an abnormality in the Echocardiogram or in the 12-lead ECG that, in the opinion of the Investigator, increases the risk of participating in the study.
7. Pulmonary function test (PFT) values of forced vital capacity (FVC) and or FEV1 < 60% predicted at the screening visit or within 6 months prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to 24 weeks
Change from Baseline in Physical Examination | Up to 24 weeks
  Physical Examination will include the assessment of body systems.
Change from Baseline in Clinical Laboratory Parameters | Up to 24 weeks
Change from Baseline in Blood Pressure | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Monique Champagne, M.Sc., Study Director — VP, Clinical Operations
Locations (2):
- Site-501, Edmonton, Alberta, Canada
- Site-202, Greifswald, Germany